CLINICAL TRIAL: NCT00057668
Title: Prevention of Behavioral Deficits in Young ADHD Children
Brief Title: Preventing Behavior Problems in Children With ADHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lehigh University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH061563 (NIH); R01MH061563 (NIH); DSIR CT-S
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2006-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Behavioral: Multi-Setting Early Intervention
Behavioral: Community Intervention

SUMMARY:
This study will determine the effectiveness of a combination of treatments in preventing behaviors that are typically associated with Attention Deficit Hyperactivity Disorder (ADHD) in young children.

DETAILED DESCRIPTION:
Participants are randomly assigned to either a Multi-Setting Early Intervention group or to a Community Intervention group. The Early Intervention group receives parent training and assessment-based behavioral and academic intervention for 1 year, followed by either a high or a low intensity maintenance intervention for an additional 18 months. The Community Intervention group members receive psychotropic medication, special education services, and monthly sessions to obtain information about child development and medical functioning for 2 years. Participants are assessed on six occasions over 4 years. Parents and teachers assess children's behavior, academic performance, and archival data, including medical and school records.

ELIGIBILITY:
Inclusion Criteria:

* Attention Deficit Hyperactivity Disorder (ADHD) diagnosis
* Preschool, nursery school, or group daycare enrollment at least 2 days per week
* Parents who can communicate in English

Exclusion Criteria:

* Plans to move out of the area in the near future
* Mental retardation, neurological damage, significant motor or physical impairments, or autism or other pervasive developmental disorder
* Inattentive ADHD or conduct disorder

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200
Dates: Start 2001-09; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Locations (1):
- Lehigh University College of Education, Bethlehem, Pennsylvania, United States